CLINICAL TRIAL: NCT07076017
Title: Effects of a 10-week Dry-land Strength and Conditioning Programme on the Start and Turn Performance of Regional- and National-level Age-group Swimmers
Brief Title: Dry-land Strength and Conditioning for Competitive Youth Swimmers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: York St John University (Other)
Collaborators: York City Baths Club (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETH2425-0466
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Swimming; Strength Training Effects; Power Training Exercise Protocols
Keywords: Non-randomised controlled trial; Youth swimmers; Strength and conditioning; Race performance

STUDY DESIGN:
Intervention Model Description: Non-randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Dry-land strength and conditioning programme
- Control group (Active Comparator)
  Interventions: Behavioral: Active control condition

INTERVENTIONS:
Behavioral: Dry-land strength and conditioning programme — Participants in the experiment group will be asked to complete two supervised gym sessions per week for 10 weeks. Each session will include a variety of plyometric and strength exercises, selected for their relevance to start and turn performance in swimming.
  Arms: Intervention group
Behavioral: Active control condition — The control group will complete their usual swimming training which comprises of several pool-based session and one land-based session each week.
  Arms: Control group

SUMMARY:
Starts and turns play an important role in swimming performance, with starts accounting for around a quarter of the total time achieved in a 50m freestyle race and have been recommended as a high priority area for improvement by York City Baths Club (YCBC). The relationship between starts and turns and plyometric and general strength training is well documented. However, few studies have explored this relationship in competitive youth swimmers. This non-randomised controlled trial will evaluate the effects of a dry-land strength and conditioning programme, when added to usual swim training, on the physical fitness and start and turn performance of regional- and national-level age-group swimmers. The study intervention will involve two supervised gym sessions per week for 10 weeks. Study outcomes will be assessed before the intervention, at the midpoint and at 1 week and 3 weeks post-intervention. The following testing will occur: Pool-based testing (50m Freestyle; a Time to 7.5m test; Turn time); Gym-based testing (Counter-movement jump; Isometric Mid-Thigh Pull; Athletic Shoulder (ASH)) The dive and turn measures will be assessed via video recordings.

ELIGIBILITY:
Inclusion Criteria:

* Member of York City Baths Club's National, Regional or Club Squads
* Age 12 to 21 years old

Exclusion Criteria:

* Parent/guardian and/or swimmer unwilling to provide written, informed consent
* Current time-loss injury
* Unable to complete 2 interventions sessions per week for 10 weeks (intervention group only)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Swim start performance | From enrolment to 3 weeks after the end of the intervention
  Time to 7.5m from a race start
Swim turn performance | From enrolment to 3 weeks after the end of the intervention
  5m turn around time during maximal effort front-crawl swimming with tumble-turn

SECONDARY OUTCOMES:
Swim race performance | From enrolment to 3 weeks after the end of the intervention
  Time to complete a maximal 50m front-crawl race
Countermovement jump performance | From enrolment to 3 weeks after the end of the intervention
  Maximum height achieved on the countermovement jump test
Lower-body strength | From enrolment to 3 weeks after the end of the intervention
  Peak force achieved on an isometric mid-thigh pull test
Shoulder strength | From enrolment to 3 weeks after the end of the intervention
  Peak force achieved in the Athletic Shoulder Test with the arm tested in the 90- and 135-degree positions

CONTACTS AND LOCATIONS:
Overall Officials: Garry Tew, PhD, Study Director — York St John University; Evelyn Wright, MSc, Principal Investigator — York St John University
Locations (1):
- York St John University, York, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided